CLINICAL TRIAL: NCT06325059
Title: Studying the Role of Renal Progenitors and Polyploid Tubular Cell Response in Glomerular and Tubular Diseases: Analysis on Renal Biopsies
Brief Title: The Role of Renal Progenitors and Polyploid Tubular Cell Response in Glomerular and Tubular Diseases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Paola Romagnani, Professor, MD, PhD, Meyer Children's Hospital IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BIO-KIDNEY
Record Dates: First submitted 2024-02-29; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Nephropathy
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Intervention Model Description: Patients affected by nephropathy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with kidney diseases undergoing renal biopsy (Experimental): Patients with kidney diseases undergoing renal biopsy for diagnostic purposes
  Interventions: Other: Study of renal progenitors

INTERVENTIONS:
Other: Study of renal progenitors — Evaluation of the role of renal progenitors in pathogenesis and mechanisms of disease progression in kidney biopsies performed for diagnostic purposes

SUMMARY:
Renal progenitors are a subset of parietal epithelial cells (PECs) localized at the urinary pole of Bowman's capsule. Experimental models of podocyte damage showed that PECs can potentially regenerate lost podocytes by migrating from Bowman's capsule to the glomerular tuft, acquiring the morphological and functional features of mature podocytes. Podocyte loss and damage, as well as the inability of PECs to replace lost podocytes, lead to glomerular scarring and chronic kidney disease (CKD) progression.

In addition, the investigators of the present study and others have recently demonstrated the existence of a specific subpopulation of tubular cells in the human kidney with a high potential for regeneration and resistance to death, thus acting as tubular progenitors. These cells are involved in tubular response to damage during acute kidney injury (AKI) trough endoreplication (polyploidization).

Kidney biopsy is the cornerstone of diagnosis in many kidney diseases leading to CKD and AKI, allowing unambiguous diagnosis in some cases and presumptive diagnosis of ongoing disease in others. Very recently, super resolution imaging techniques proved to maintain current diagnostic standards while allowing to study morphological features of pathophysiological mechanisms of glomerular and tubular diseases.

The rationale of this project is to study the role of renal progenitors (PECs and tubular progenitors) in the pathogenesis of CKD and AKI trough super resolution imaging applied to human renal biopsies, to the aim of identifying relevant connections with clinical data and markers of damage and/or disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients with glomerular diseases undergoing renal biopsy (e.g., rapidly progressive glomerulonephritis, minimal change disease, focal segmental glomerulosclerosis, diabetic nephropathy, lupus nephritis, membranous nephropathy, IgA nephropathy, etc)
* Patients with AKI, regardless of the nature of the damage (septal, ischemic, toxic, or unknown).
* Signed informed consent form

Exclusion Criteria:

* Sample insufficient and/or unavailable

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2023-03-22 (Actual); Primary Completion 2047-03-22 (Estimated); Study Completion 2047-11-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the role of renal progenitors in the progression of glomerular diseases | Clinical data will be collected at enrollment (kidney biopsy) and at 3, 6 and 12 months from enrollment, then annually until the end of the study (up to 9 years)
  The presence renal progenitors will be assessed by immunofluorescence and confocal microscopy on histological sections from renal biopsy performed for diagnostic purposes.
  The following features will be assessed and correlated with clinical parameters of renal function:
  * number of renal progenitors (CD133+CD24+CD106+ cells/section);
  * number of podocyte progenitors (CD133+WT1+, CD24+synaptopodin, CD24+podocin+ cells/section);
  * number of activated progenitors in the Bowman's capsule (CD133+SFN+/section)
  * quantitative and semiqualitative analysis of the slit diaphragm
  * presence and characterization of immune complexes

SECONDARY OUTCOMES:
Evaluation of the role of tubular endoreplication in mechanisms of acute kidney injury (AKI) | Clinical data will be collected at enrollment (kidney biopsy) and at 3, 6 and 12 months from enrollment, then annually until the end of the study (up to 9 years)
  The presence of tubular progenitors will be assessed by immunofluorescence and confocal microscopy evaluation on histological sections from renal biopsy performed for diagnostic purposes. The presence of polyploid tubular cells will be assessed using specific markers.
  In particular, the following features will be assessed:
  * number of tubular progenitors (CD133+CD24+CD106- cells) over the total of tubular cells (phaIIoidin+, AQP1+, THP+, AQP2+ cells);
  * number of Ki-67+ or PCNA+ over the total of tubular cells (%);
  * number of polyploid tubular cells (CDK4+ or CDT1+ and p-H3+) over the total of tubular cells;
Evaluation of the role of tubular endoreplication in mechanisms of acute kidney injury (AKI) trough DNA and RNA analysis | Clinical data will be collected at enrollment (kidney biopsy) and at 3, 6 and 12 months from enrollment, then annually until the end of the study (up to 9 years)
  The presence of tubular progenitors will be assessed by immunofluorescence and confocal microscopy evaluation on histological sections from renal biopsy performed for diagnostic purposes. The presence of polyploid tubular cells will be assessed using specific markers, in particular:
  * DNA content (fluorescence intensity of Picogreen/YAP1 staining);
  * RNA expression of polyploidy markers (TMSB10, SEMA5a, VCAM1, BIRC5, AKT, E2F7, E2F8, CDK1, CCNB1)

CONTACTS AND LOCATIONS:
Locations (1):
- Meyer Children's Hospital IRCCS, Florence, Italy

IPD SHARING:
Plan to Share IPD: No